CLINICAL TRIAL: NCT00809640
Title: Active Management for Low Back Pain Taught to 6 to 8 Year Old Schoolchildren
Brief Title: Active Management for Low Back Pain for 6 to 8 Year Old Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kovacs Foundation (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FK 27
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Low Back Pain
Keywords: low back pain; prevention; schoolchildren; education campaign
MeSH Terms: conditions — Low Back Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The intervention group will receive prevention of low back pain education through a Back Comic-Book, and their beliefs/knowledge will be tested twice after intervention.
  Interventions: Behavioral: Education (Back Comic-Book)
- 2 (No Intervention): The control group will receive no intervention, and their beliefs/knowledge on low back pain will be tested twice after the first assessment.

INTERVENTIONS:
Behavioral: Education (Back Comic-Book) — Through the Back Comic-Book the schoolchildren are taught prevention methods for low back pain.
  Arms: 1

SUMMARY:
The objective is to assess the effectiveness of a prevention campaign promoting active management in shifting beliefs in 6 to 8 year old schoolchildren. Subjects will be taken from a random sample of schools in Majorca, Spain: private, public and concerted. A 10 item questionnaire will be given to all children in that age group, to be answered in class on days 1, 14 and 97. Schools will be randomly assigned to the study and control groups. In the study group the students will get a Back Comic-Book (promotes active management) after the first assessment. The control group will have no other intervention than the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Students in randomly selected private, public and concerted Majorca schools
* Must be present in class on day of intervention and assessments

Exclusion Criteria:

* Absent from class on day of intervention and assessments

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the effectiveness of a prevention campaign promoting active management of low back pain in shifting beliefs in 6 to 8 year old schoolchildren. | 4 months
Assessment of the effectiveness of a prevention campaign promoting active management on low back pain in 6 to 8 year old schoolchildren. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Mario Gestoso, MD, Principal Investigator — Kovacs Foundation,Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain